CLINICAL TRIAL: NCT03758690
Title: Efficacy of Abdominal Treatment With High-Intensity Focused Electromagnetic (HIFEM) Field Device in Women After Childbirth
Brief Title: High-Intensity Focused Electromagnetic (HIFEM) Field Device in Women After Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-After Childbirth
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Muscle Tone Increased
MeSH Terms: conditions — Muscle Hypertonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Treatment with the investigational device - High-Intensity Focused Electromagnetic (HIFEM) Field Device
  Interventions: Device: High-Intensity Focused Electromagnetic (HIFEM) Field Device

INTERVENTIONS:
Device: High-Intensity Focused Electromagnetic (HIFEM) Field Device — The High-Intensity Focused Electromagnetic (HIFEM) Field device will be applied.

SUMMARY:
Evaluation of use of the High-Intensity Focused Electromagnetic (HIFEM) Field Device in women after childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Non-breastfeeding women 3-36 months after childbirth
* Voluntarily signed informed consent form
* BMI ≤ 30 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Implanted defibrillators, implanted neurostimulators
* Electronic implants
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Application in the head area
* Application in the heart area
* Malignant tumor
* Fever
* Pregnancy
* Breastfeeding
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over areas of the skin which lack normal sensation
* Scars, open lesions and wounds at the treatment area
* Unrepaired abdominal hernia
* Patients after Cesarean section delivery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the device for abdominal toning according to MRI images | 7 months
  Evaluation of MRI images before and after the therapy procedure.
Effectiveness of the device for abdominal toning according to waist circumference measurements | 7 months
  Evaluation of waist circumference measurements (in centimeters).

SECONDARY OUTCOMES:
Subject's satisfaction with study treatment: Questionnaire | 7 months
  Subject's satisfaction with the therapy results evaluated through the Subject Satisfaction Questionnaire. The 7-point Likert scale Subject Satisfaction Questionnaire will be used for an analysis of the subject's opinion of the therapy results.
Determination of side effects and adverse events (AE) associated with the study device. | 7 months
  The occurrence of side effects and adverse events will be followed throughout the whole study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois